CLINICAL TRIAL: NCT06353425
Title: Multi-country Survey on Violence Against Women Among Reproductive-aged Women
Brief Title: Multi-country Survey on Violence Against Women Among Women
Status: Not yet recruiting | Type: Observational
Sponsor: Chulalongkorn University (Other)
Collaborators: Asia and Oceania Federation of Obstetrics and Gynaecology (Unknown)
Responsible Party: Principal Investigator, Unnop Jaisamrarn, Professor, Chulalongkorn University
Other Study IDs: 0562/66
Record Dates: First submitted 2024-03-19; First posted 2024-04-09 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Violence Against Women
Keywords: reproductive-aged women; violence against women; gender-based violence; knowledge; attitude; practice
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Reproductive aged women: Reproductive aged women in Asia and Oceania countries

SUMMARY:
The goal of this observational study is to explore and learn about violence against women (VAW) among reproductive-aged women in Asia and Oceania countries. The main questions it aims to answer are:

* pattern and prevalence of VAW among reproductive-aged women
* knowledge, attitude, and practice (KAP) towards VAW among reproductive-aged women
* the need of support services for VAW among reproductive-aged women

Participants will be ever-partnered women aged 15-49 years. The definition of "ever-partnered women" included women who have current and former husbands; current and former cohabiting; or non-cohabiting male intimate partners.

DETAILED DESCRIPTION:
Violence against women (VAW) is a global issue that threatens women's physical and emotional wellbeing, and impacts women worldwide, regardless of age, race, ethnicity, or nationality. This survey aims to investigate 1) the pattern and prevalence of VAW among reproductive-aged women; 2) the knowledge, attitude, and practice (KAP) towards VAW among reproductive-aged women; and 3) the need of support services for VAW among reproductive-aged women.

This multinational, hospital-based, cross-sectional study will be carried out in Asia and Oceania countries. We will select the Obstetrics and Gynecology Outpatient Department or Women Health Unit in each nation. Minimum of 400 female citizen in each country will be recruited if they are aged 15-49 years, ever-partnered women, and agree to finish the questionnaire.

The questionnaire, developed in English with inputs from literature and experts, comprises four sections: 1) basic participant characteristics, 2) patterns and prevalence of violence, 3) knowledge, attitudes, and practices towards violence, and 4) the need for support services. A pilot study will validate and translate the questionnaire into the target languages, ensuring content relevance and sensitivity to the target culture through forward and backward translation processes. The reliability of the questionnaire will be assessed using Cronbach's alpha.

Data collection involves preparatory steps such as developing a training manual for interviewers, addressing potential issues, and advertising the survey. Central investigators will monitor the data collection process, with data collected through self-administered questionnaires. The use of REDCap software aims to manage surveys efficiently and prevent multiple participations. A paper-based questionnaire could be used in some areas when necessary.

ELIGIBILITY:
Inclusion Criteria:

* ever-partnered women
* aged 15-49 years

The definition of "ever-partnered women" included women who have current and former husbands; current and former cohabiting; or non-cohabiting male intimate partners.

Exclusion Criteria:

* declined to participate
* dropped out midway

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Women in Asia and Oceania countries, who register at the Obstetrics and Gynecology Outpatient Department or Women Health Unit. Participant's biological sex should be female.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
prevalence of violence against women | through study completion, an average of 1 year
  using questionnaire to explore the prevalence of various forms of violence against women
KAP towards violence against women | through study completion, an average of 1 year
  using questionnaire to explore knowledge, attitude, and practice towards violence against women

SECONDARY OUTCOMES:
need of support services for violence against women | through study completion, an average of 1 year
  using questionnaire to identify the need of support services for violence against women among reproductive-aged women

CONTACTS AND LOCATIONS:
Overall Officials: Unnop Jaisamrarn, MD,MHS, Principal Investigator — Chulalongkorn University

IPD SHARING:
Plan to Share IPD: Undecided
Since this will be a multinational survey, we will decide after discussing about this issue with investigators of each country.